CLINICAL TRIAL: NCT02791451
Title: Open-Label Prospective Study of Predicting Exacerbation of Chronic Obstructive Pulmonary Disease (COPD) With Wireless Telemonitoring of Respiratory Rate, Heart Rate and Sleep
Brief Title: Predicting Exacerbation of COPD With Wireless Telemonitoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The device did not provide sufficient quality of data
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COPD_BCG
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: COPD
Keywords: COPD; telemonitoring; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemonitoring (Experimental): Exacerbation of COPD with wireless telemonitoring of respiratory rate, heart rate and sleep.
  Interventions: Device: telemonitoring

INTERVENTIONS:
Device: telemonitoring — To predict exacerbation of COPD with wireless telemonitoring

SUMMARY:
This is an open-label single-center 6-month prospective clinical trial predicting exacerbation of COPD with wireless telemonitoring of respiratory rate, heart rate and sleep in patients admitted to the pulmonary ward of the Turku University Hospital due to acute exacerbation of COPD.

DETAILED DESCRIPTION:
A bed sensor based on ballistocardiogram (BCG) will be used to wireless telemonitoring of respiratory rate, heart rate and sleep for six months after an acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients treated due to acute exacerbation of COPD at the pulmonary wards of the Turku University Hospital

Exclusion Criteria:

* Those sleeping with a bed partner and not having separate mattresses
* Patients with pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time window to detect acute exacerbation of COPD | Six months
  Time window to detect acute exacerbation of COPD

IPD SHARING:
Plan to Share IPD: No